CLINICAL TRIAL: NCT04615806
Title: The Value of Lymph Node Dissection of Indocyanine Green-guided Near-infrared Fluorescent Imaging in Video-assisted Thoracoscope Radical Esophagectomy
Brief Title: The Value of Lymph Node Dissection of Indocyanine Green-guided Near-infrared Fluorescent Imaging in Esophagectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICG-NIR UNION
Record Dates: First submitted 2020-10-27; First posted 2020-11-04 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Esophageal Cancer; Indocyanine Green
Keywords: Esophageal Cancer; Indocyanine Green; the lymph node markers
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Indocyanine Green; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIR-ICG (Experimental): After positioning,Indocyanine green（ICG） dye (Yichuang Pharmaceutical, Liaoning, China) stored at a dose of 25 mg in a small bottle was diluted with 5 ml sterile water. Then, 2 ml of this solution was added to 8 ml sterile water in a dis-posable dressing bowl, resulting in a final concentration of 1.25 mg/ml.
  Interventions: Drug: Indocyanine green solution
- Control (No Intervention): This group of patients received only conventional radical resection of esophageal cancer without Indocyanine green injection.

INTERVENTIONS:
Drug: Indocyanine green solution — ICG solution was endoscopically injected into the esophageal submucosa at the four quadrants around the tumor.
  Other Names: Indocyanine Green for Injection
  Arms: NIR-ICG

SUMMARY:
Indocyanine green (ICG) has been recently introduced in clinical practice as a fuorescent tracer. Lymphadenectomy is particularly challenging in esophageal cancer surgery, owing to the complex anatomical drainage.Therefore, the purpose of this study was to explore whether the NIR-ICG imaging system could accurately assess the lymph node markers during radical resection of esophageal cancer.

DETAILED DESCRIPTION:
This study will be accepted in esophageal cancer patients with Radical Esophag-ectomy as the research object.We will divide them into two groups: experimental group for injection of indocyanine green group and control group for injectable in-docyanine green group.We will compare with the accuracy,false positive rate and false negative rate,sensitivity, specificity and related indicators of intraoperative lymph node cleaning,in order to explore the common position of esophageal cancer sentinel lymph node,guidance of esophageal cancer lymph node cleaning thoroughly.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: 18-75 years old, male and female unlimited;
2. Preoperative biopsy was pathologically diagnosed as esophageal squamous cell carcinoma;
3. Preoperative combination with neoadjuvant chemoradiotherapy;
4. Surgical resection of esophageal carcinoma under endoscopic selection and intraoperative anastomosis;
5. Heart, lung, liver and kidney functions can tolerate operation;
6. Patients and their family members can understand and are willing to participate in this clinical study and sign the informed consent.

Exclusion Criteria:

1. Allergic to ICG or iodine;
2. Patients with a history of chest surgery or thoracic lymph node dissection;
3. Patients needing emergency surgery;
4. Patients whose tumors involve neighboring organs and need to be removed by combining organs;
5. Patients with tumor recurrence or distant metastasis;
6. Patients who had participated in or were participating in other clinical trials within the previous 4 weeks were included;
7. A history of serious mental illness;
8. Pregnant or lactating women;
9. Patients with other conditions considered by the researcher should not participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy rate of lymph node dissection | 1 week after operation
  Accuracy rate of lymph node dissection of each arm（according to postoperative pathology）
False positive rate of lymph node dissection | 1 week after operation
  False positive rate of lymph node dissectionof each arm（according to postoperative pathology）
False negative rate of lymph node dissection | 1 week after operation
  False negative rate of lymph node dissection of each arm（according to postoperative pathology）
Sensitivity and specificity of lymph node dissection | 1 week after operation
  Sensitivity and specificity of lymph node dissection of each arm（according to postoperative pathology）

SECONDARY OUTCOMES:
The mapping of sentinel lymph nodes in esophageal cancer | 1 week after operation
  The mapping of sentinel lymph nodes in esophageal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chen, MD, Study Director — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Du J, Zeng T, Zhang S, Chen M, Huang G, Xu C, Xu G, Ni C, Hong R, Zheng W, Chen C, Zheng B. Comparison of indocyanine green-near-infrared fluorescence guided and traditional mediastinal lymphadenectomy during radical esophagectomy: A randomized controlled trial. Surgery. 2024 Feb;175(2):347-352. doi: 10.1016/j.surg.2023.10.007. Epub 2023 Nov 26. PMID 38012899
- [Derived] Du J, Xu G, Yang Z, Zheng B, Chen C. Pericancerous lymph node imaging with indocyanine green-guided near-infrared fluorescence in radical esophagectomy: Protocol for a single-center, prospective, randomized controlled clinical trial. Thorac Cancer. 2022 Aug;13(15):2283-2287. doi: 10.1111/1759-7714.14548. Epub 2022 Jun 29. PMID 35770339